CLINICAL TRIAL: NCT01467349
Title: Efficacy of Raltegravir in a Large Urban HIV Clinic Population in Milan (Efficacy of Raltegravir in a Large Urban HIV Clinic Setting)
Brief Title: Efficacy of Raltegravir in a Large Urban HIV Clinical Population in Milan
Acronym: Real-Life
Status: Completed | Type: Observational
Sponsor: Università Vita-Salute San Raffaele (Other)
Collaborators: Ospedale San Raffaele (Other)
Responsible Party: Principal Investigator, Elisabetta Carini, Professor Massimo Clementi, Università Vita-Salute San Raffaele
Other Study IDs: Real-Life Study; Real-Life (Other Grant/Funding Number: Merck Sharp & Dohme)
Record Dates: First submitted 2011-11-03; First posted 2011-11-08 (Estimated); Last update posted 2013-02-11 (Estimated); Status verified 2013-02

CONDITIONS: HIV Infections
Keywords: Raltegravir; efficacy; safety; raltegravir-containing regimens; HIV urban clinic setting
MeSH Terms: conditions — HIV Infections

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Raltegravir group: This study will include subjects who received raltegravir and were previously exposed to NRTIs, NNRTIs, PIs, regardless of the stage of HIV disease at the start of the treatment.
  A control group will be used for the evaluation of the primary and secondary objectives in comparison to patients treated with raltegravir (study patients). The control group will be constituted by subjects who never received raltegravir, matched (in a ratio 1:3) with the study subjects by gender, age (± 3 years), CD4+ cells counts (± 50 cells) and HCV co-infection status yes/no). For control patients, the last antiretroviral regimen prescribed will be considered.

SUMMARY:
This will be a retrospective analysis of efficacy, safety and tolerability of raltegravir as part of an optimized therapy in a clinical setting.

Follow-up is calculated from the treatment initiation (with or without raltegravir) up to the date of discontinuation of the considered regimen or the date of last visit or the date of lost to follow-up, whichever came first.

The Aim of the study is to evaluate the efficacy and safety of raltegravir-containing regimens in a urban clinic setting.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who received raltegravir and were previously exposed to NRTIs, NNRTIs, PIs, regardless of the stage of HIV disease at the start of the treatment.

Exclusion Criteria:

* None

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study will include subjects who received raltegravir and were previously exposed to NRTIs, NNRTIs, PIs, regardless of the stage of HIV disease at the start of the treatment.
  A control group will be used for the evaluation of the primary and secondary objectives in comparison to patients treated with raltegravir (study patients). The control group will be constituted by subjects who never received raltegravir, matched (in a ratio 1:3) with the study subjects by gender, age (± 3 years), CD4+ cells counts (± 50 cells) and HCV co-infection status yes/no). For control patients, the last antiretroviral regimen prescribed will be considered.
Sampling Method: Probability Sample
Enrollment: 400 (Actual)
Dates: Start 2011-12; Primary Completion 2012-10 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Real-Life | baseline and week 48
  Primary endpoint is the proportion of patients with HIV-1 RNA<50 copies/ml at weeks 48 after treatment initiation (baseline).

SECONDARY OUTCOMES:
Real-Life | baseline and week 48
  Secondary endpoints are:
  * Proportion of patients with HIV-1 RNA<50 copies/ml at the end of the treatment/last available visit
  * Proportion of patients with HIV-1 RNA<400 copies/ml at week 48
  * Increase in absolute CD4 cell count from baseline
  * Frequency of side effects associated with raltegravir treatment
  * Frequency of reasons for starting/stopping raltegravir treatment

CONTACTS AND LOCATIONS:
Overall Officials: Massimo Clementi, Prof., Principal Investigator — Università Vita-Salute
Locations (1):
- Infectious Diseases Department, Milan, Milan, Italy

REFERENCES:
- [Background] Steigbigel RT, Cooper DA, Kumar PN, Eron JE, Schechter M, Markowitz M, Loutfy MR, Lennox JL, Gatell JM, Rockstroh JK, Katlama C, Yeni P, Lazzarin A, Clotet B, Zhao J, Chen J, Ryan DM, Rhodes RR, Killar JA, Gilde LR, Strohmaier KM, Meibohm AR, Miller MD, Hazuda DJ, Nessly ML, DiNubile MJ, Isaacs RD, Nguyen BY, Teppler H; BENCHMRK Study Teams. Raltegravir with optimized background therapy for resistant HIV-1 infection. N Engl J Med. 2008 Jul 24;359(4):339-54. doi: 10.1056/NEJMoa0708975. PMID 18650512
- [Background] Lennox JL, Dejesus E, Berger DS, Lazzarin A, Pollard RB, Ramalho Madruga JV, Zhao J, Wan H, Gilbert CL, Teppler H, Rodgers AJ, Barnard RJ, Miller MD, Dinubile MJ, Nguyen BY, Leavitt R, Sklar P; STARTMRK Investigators. Raltegravir versus Efavirenz regimens in treatment-naive HIV-1-infected patients: 96-week efficacy, durability, subgroup, safety, and metabolic analyses. J Acquir Immune Defic Syndr. 2010 Sep;55(1):39-48. doi: 10.1097/QAI.0b013e3181da1287. PMID 20404738